CLINICAL TRIAL: NCT03037788
Title: Pharmacokinetics, Local and Systemic Tolerability and Local Efficacy of Ascending Concentrations of Glycopyrronium Bromide (GPB) in a Topical Formulation in a Placebo Controlled, Double Blind Study in Subjects With Axillary Hyperhidrosis
Brief Title: Investigation of Ascending Concentrations of Glycopyrronium Bromide (GPB) in a Topical Formulation in Subjects With Axillary Hyperhidrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. August Wolff GmbH & Co. KG Arzneimittel (Industry)
Collaborators: Nuvisan GmbH (Unknown); FGK Clinical Research GmbH (Industry); Charles River Biopharmaceutical Services GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Hyp-02/2015; 2015-005570-38 (EudraCT Number)
Record Dates: First submitted 2016-12-21; First posted 2017-01-31 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2017-07

CONDITIONS: Primary Axillary Hyperhidrosis
Keywords: Excessive sweating
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- WO3979 (Experimental): Formulation containing WO3979 for topical application
  Interventions: Drug: WO3979
- WO3970 (Experimental): Formulation containing WO3970 for topical application
  Interventions: Drug: WO3970
- WO3992 (Experimental): Formulation containing WO3992 for topical application
  Interventions: Drug: WO3992
- Placebo of WO3988 (Placebo Comparator): Formulation containing Placebo of WO3988 for topical application
  Interventions: Drug: Placebo (WO3988)

INTERVENTIONS:
Drug: WO3979 — Application of cream to each axilla
  Arms: WO3979
Drug: WO3970 — Application of cream to each axilla
  Arms: WO3970
Drug: WO3992 — Application of cream to each axilla
  Arms: WO3992
Drug: Placebo (WO3988) — Application of cream to each axilla
  Arms: Placebo of WO3988

SUMMARY:
The aim of the study is to assess the safety, tolerability, pharmacokinetics (PK) and efficacy of escalating concentrations of GPB in subjects with axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe primary axillary hyperhidrosis whose HDSS score is 2, 3 or 4
* At least 50 mg in males or 25 mg in females of spontaneous resting axillary sweat production in one axilla measured gravimetrically at room temperature/humidity (about 25°C / 20-50%) over a period of 5 minutes.
* Male and female subjects in the age of 18 to 65 years at the time of informed consent and a body mass index (BMI) of 18-32 kg/m2.
* Corrected QT (QTc) ≤450 msec, or QTc <480 msec in subjects with bundle branch block.
* Able to comply with protocol requirements, including overnight stays, blood sample collections as defined in the protocol subjects.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Known allergy to any of the components in the investigational product.
* Hypersensitivity against glycopyrrolate
* Secondary hyperhidrosis, for example, hyperhidrosis that is secondary to other underlying diseases including hyperthyroidism, lymphoma and malaria, climacteric hyperhidrosis.
* Previous surgical treatment of hyperhidrosis including sympathectomy, surgical debulking of the sweat glands, subcutaneous tissue curettage and ultrasonic surgery.
* Botulinum toxin treatment in the prior 9 months.
* Present or history of neuromuscular disease.
* Angle closure glaucoma or its precipitation (narrow angle).
* Mycotic, other skin infections and other dermal disorder including infection at anticipated application sites in either axilla.
* Significant cardiac arrhythmia such as tachycardiac atrial fibrillation and very frequent extrasystoles.
* Subject with diabetes mellitus.
* Subjects with ileus, gastrointestinal stenosis, pronounced chronic inflammatory bowel disease, toxic megacolon.
* Subjects with epilepsy.
* Use of antiperspirants containing aluminium chloride and deodorants, any oral herbal medicine treatments or any other topical treatments for hyperhidrosis within 7 days prior to study treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety assessed through adverse events and local skin reactions | 3 weeks

SECONDARY OUTCOMES:
Gravimetric measurement of sweat production | 3 weeks
Dermatology Life Quality Index (DLQI) | 3 weeks
Hyperhidrosis Disease Severity Scale (HDSS) | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Christoph Abels, MD, PhD, Study Director — Dr. August Wolff GmbH & Co. KG Arzneimittel; Horst Jürgen Heuer, MD, Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No